CLINICAL TRIAL: NCT04175548
Title: Cut-out of the Cervical Screw on Pertrochanteric Fractures: Retrospective Analysis of 12 Cases
Brief Title: Cut-out of the Cervical Screw on Pertrochanteric Fractures
Status: Completed | Type: Observational
Sponsor: Tamas Illes (Other)
Responsible Party: Sponsor-Investigator, Tamas Illes, Head of Orthopedic Surgery Department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Lahsika
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Pertrochanteric Fracture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surgery for a pertrochanteric fracture: Patients having had surgery for a pertrochanteric fracture at the CHU Brugmann Hospital between January 2013 and May 2019.
  Interventions: Other: Data extraction from medical files

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
Pertrochanteric fractures are a highly relevant topic not only because of the high frequency or age of the population concerned, but also because of comorbidity (osteoporosis, malnutrition, decreased physical activity, decreased visual acuity, neurological deficits, asthenia, disorders of the equilibrium and impaired reflexes) and the mortality associated with this type of fractures.

The cut-out of the cervical screw is a mechanical complication common to different means of osteosynthesis of pertrochanteric fractures, this complication significantly increases the morbidity.

From January 2013 to May 2019, out of a total of 340 patients having had surgery for pertrochanteric fracture, 12 cases of cervical screw cut-out were recorded within the Brugmann University Hospital. The average follow-up after surgery was 18 months.

This study analyses different parameters and their link with cervical screw cut-outs, and compares the results with the ones published in the scientific literature.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted for a pertrochanteric and subtrochanteric fracture of the femur treated by cerebrospinal nailing with all the methods of fixation of the head (blade or screw) and who evolved to a cut-out of the cervical screw.

Exclusion Criteria:

* Fractures treated by open osteosynthesis
* Fractures operated with good radiological outcome
* Incomplete or non useable medical files

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted for a pertrochanteric and subtrochanteric fracture of the femur treated by cerebrospinal nailing with all the methods of fixation of the head (blade or screw) and who evolved to a cut-out of the cervical screw.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Ender Classification | 5 minutes
  Ender classification of the fracture. I: stable basal-cervical fracture. II: stable pertrochanteric fracture. III: unstable intertrochanteric fracture. IV: unstable subtrochanteric fracture. V: unstable trochantero-diaphyseal fracture
Bone quality | 5 minutes
  Presence of osteoporosis or pathologies inside the bone (yes/no)
Type of osteosynthesis | 5 minutes
  Material used. Choice between: short/long gamma nail, long/short PFNA nail, long/short Affixus nail
Correct positioning of the screw | 5 minutes
  Correct positioning of the screw on radiological images (yes/no)
Delay between fracture and screw cut-off | up to 18 months
  Delay between fracture and screw cut-off
Tip Apex Distance (TAD) | 5 minutes
  TAD is a measure of how close the tip of the lag screw lies to the femoral apex.
Parker ratio | 5 minutes
  This method involves recording the superior, inferior, anterior and posterior borders of the femoral head. The ratio is calculated in both the AP and lateral views to give a value within a range of 0 to 100 for each view. In the AP view, 0 is considered to be the most inferior screw placement and 100 is considered to be the most superior pin placement. In the lateral view, 0 is considered to be the most posterior screw placement and 100 is considered to be the most anterior pin placement.
Age | 5 minutes
  Age of the patient
Sex | 5 minutes
  Sex of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Lahsika, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No